CLINICAL TRIAL: NCT04249856
Title: Does Dynamic Spectral Imaging (DSI) Colposcopy Improve the Diagnostics of Cervical Dysplasia Compared to Standard Colposcopy
Brief Title: Colposcopy and Dynamic Spectral Imaging (DSI)
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University of Aarhus (Other)
Responsible Party: Sponsor
Other Study IDs: DSIcolposcopy_DK
Record Dates: First submitted 2020-01-23; First posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2019-12

CONDITIONS: Cervical Dysplasia; Cervical Disease; Cervical Lesion; Cervix Cancer; Cervical Cancer; Cervical Neoplasm
Keywords: Colposcopy; Dynamic Spectral Imaging, DySIS; Colposcopy Directed Biopsy
MeSH Terms: conditions — Uterine Cervical Dysplasia; Uterine Cervical Diseases; Uterine Cervical Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Cervical punch biopsies
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

GROUPS / COHORTS (1):
- Women examined by colposcopy: Women referred to colposcopy at our facilities who met inclusion criteria
  Interventions: Diagnostic Test: Dynamic Spectral Imaging (DYSIS)

INTERVENTIONS:
Diagnostic Test: Dynamic Spectral Imaging (DYSIS) — Women who have a colposcopy exam performed at Randers Regional Hospital were examined by Dynamic Spectral Imaging colposcopy (DYSIS)

SUMMARY:
This study evaluates the Dynamic Spectral Imaging (DSI) Colposcope (DySIS) in it's ability to diagnose cervical dysplasia. Half of participants with be examined by the DySIS colposcope, there the other half will be examined by standard colposcopy.

DETAILED DESCRIPTION:
Colposcopy has been shown to be a subjective exam, and is dependant on the colposcopists. Sensitivity for colposcopy has been shown to be as low as 50%.

To improve this, different adjunctive technologies have been introduced to add a more objective approach to the colposcopy exam. One of these devices is the DySIS colposcope, which measures the aceto-white reaction that may occur on the cervix uteri after the application of acetic-acid. The device provides the examiner with a colour-coded map indicating areas of interest. Studies have shown promising results indicating that using this device together with the colposcopists own interpretation of the cervix uteri can potentially lead to an increase in the performance of the colposcopy exam.

In Denmark all women referred for colposcopy have 4 biopsies taken, according to the Danish national guidelines.

In our study these 4 biopsies are as following:

1. The area the colposcopists views as the worst before the DSI-map is seen. Colposcopy-Directed Biopsy (CDB)
2. The area indicated as the worst by the DSI-map (DSI-directed biopsy)
3. additional biopsy
4. additional biopsy All biopsies are placed in separate containers and analysed separately by specialized pathologists.

ELIGIBILITY:
Inclusion Criteria:

* Referred for colposcopy due to a cervical smear test of Atypical Squamous Cells of Undetermined Significance (ASCUS), low-grade intraepithelial lesion (LSIL), atypical squamous cells, cannot exclude a high-grade lesion (ASC-H), high-grade intraepithelial lesion (HSIL), Atypical glandular cells (ACG) or carcinoma in situ (CIS)
* Referred for colposcopy due to follow-up of previously diagnosed CIN (If there has been a minimum of 6 months since previous cervical biopsies)

Exclusion Criteria:

* Cervical biopsies taken within the last 6 months
* Previous cone procedure
* Currently pregnant
* Pregnant within the last 6 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Female
Study Population: All women above the age of 18 who are referred for colposcopy due to an abnormal cervical smear (ASCUS, LSIL, ASC-H, HSIL, ACG or CIS) or as follow up to previously diagnosed CIN. The women cannot be included if they have had cervical biopsies taken within the last 6 months, have previously had a cone biopsy taken, are currently pregnant or have been pregnant within the last 3 months.
Sampling Method: Probability Sample
Enrollment: 3000 (Estimated)
Dates: Start 2017-02-01 (Actual); Primary Completion 2020-06-01 (Estimated); Study Completion 2020-10-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of women found with a histological diagnosis of Cervical Intraepithelial Neoplasia grade 2 or worse (CIN2+) in colposcopy-directed biopsy (CDB) | when the histological report is available - typically 4 weeks after the biopsy was taken.
  The proportion of women who are found with a histological CIN2+ diagnosis in the cervical punch biopsy from the area chosen by the colposcopist before the DSI-map became visible (will be referred to as the Colposcopy directed biopsy (CDB)).
  The diagnosis of the biopsy will be recorded when the histological report is available.
  Further treatment needs for the patient will be based on the national clinical guidelines on cervical dysplasia.
Proportion of women found with a histological diagnosis of CIN2 or worse in DSI-directed biopsies | when the histological report is available - typically 4 weeks after the biopsy was taken.
  The proportion of women who are found with a histological CIN2+ diagnosis in cervical punch biopsy taken from the worst area indicated by the DSI-map (referred to as the DSI-directed biopsy) The diagnosis of the biopsy will be recorded when the histological report is available.
  Further treatment needs for the patient will be based on the national clinical guidelines on cervical dysplasia.
Proportion of women found with a histological diagnosis of CIN2 or worse in 2 additional random biopsies | when the histological report is available - typically 4 weeks after the biopsy was taken.
  The amount of women who are found with a histological CIN2+ diagnosis in cervical punch biopsies taken from 2 additional areas besides the CDB and the DSI-directed areas.
  The diagnosis of the biopsy will be recorded when the histological report is available.
  Further treatment needs for the patient will be based on the national clinical guidelines on cervical dysplasia.

SECONDARY OUTCOMES:
Concordance of cervical punch biopsies and cone biopsy | When both histological reports were available these were compared.
  Comparing the histological diagnosis of the cervical punch biopsies to the cone biopsy, in women who are referred for conization based on the histological outcome of the colposcopy procedure.

CONTACTS AND LOCATIONS:
Overall Officials: Berit B Booth, MD, Principal Investigator — University of Aarhus; Pinar Bor, MD, PhD, Study Chair — Randers Regional Hospital; Lone K Petersen, MD, Med.Sc.D., Study Chair — Odense University Hospital; Jan Blaakaer, MD, Med.Sc.D., Study Chair — Odense University Hospital; Katja Dahl, MD, PhD, Study Chair — Aarhus University Hospital
Locations (4):
- Denmark (4):
  - Randers Regional Hospital, Randers, Danmark
  - Aalborg University Hospital, Aalborg
  - Private Gynaecology Clinic, Aarhus
  - Horsens Regional Hospital, Horsens

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Jespersen MM, Booth BB, Petersen LK. Can biopsies be omitted after normal colposcopy in women referred with low-grade cervical cytology? A prospective cohort study. BMC Womens Health. 2021 Nov 19;21(1):394. doi: 10.1186/s12905-021-01537-5. PMID 34798899
- [Derived] Booth BB, Petersen LK, Blaakaer J, Johansen T, Mertz H, Dahl K, Bor P. Can the dynamic spectral imaging (DSI) color map improve colposcopy examination for precancerous cervical lesions? A prospective evaluation of the DSI color map in a multi-biopsy clinical setting. BMC Womens Health. 2021 Jan 12;21(1):21. doi: 10.1186/s12905-020-01169-1. PMID 33435974